CLINICAL TRIAL: NCT03052621
Title: Revisiting Omental Transposition in Locally Advance and Locally Recurrent Breast Cancer
Status: Completed | Type: Observational
Sponsor: Queen Sirikit Centre for Breast Cancer (Other)
Responsible Party: Principal Investigator, Sikrit Denariyakoon, Doctor, Queen Sirikit Centre for Breast Cancer
Other Study IDs: 635/59
Record Dates: First submitted 2017-01-05; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Survival Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Curative group: Locally advance breast cancer and locally recurrent breast cancer without metastasis underwent omental transposition
  Interventions: Procedure: Omental transposition
- Palliative group: Locally advance breast cancer and locally recurrent breast cancer with metastasis underwent omental transposition
  Interventions: Procedure: Omental transposition

INTERVENTIONS:
Procedure: Omental transposition — Harvesting the omentum to cover irradiated defects of breast cancer
  Other Names: Omental graft

SUMMARY:
Locally advance breast cancer and extensive locoregional recurrence are still considered as complexity of reconstruction. Although previous studies concluded that omental transposition was considerably indicated in poor vascularity in irradiated tissue, secondary infection and large defect become the obstacles of local tissue flaps. While some centres showed the excellent healing of omental transposition. Meanwhile, many studies showed the preferable outcome in escalating radiotherapy in term of locoregional control. In the investigators' institute, omental transposition in breast cancer has been developed for twenty years. The only institute in Thailand enhanced using this procedure in order to closure of large primary breast cancer and chest wall recurrence. This procedure is undertaken by single surgeon (Dr. K.J.). The investigators' protocol of omental transposition is including preoperative chemotherapy, preoperative accelerated radiation up to 80 Gy, approval of breast cancer centre committee, and meticulous wound care including vacuum assisted wound dressing, non-adhesive dressing. As a result, survival time could be improved.

ELIGIBILITY:
Inclusion Criteria:

* The patients with omental transposition operation within King Chulalongkorn Memorial Hospital
* More than 18 years of age

Exclusion Criteria:

* The patients with refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with locally advance or locally recurrent breast cancer that aggressive chemoradiation needed.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 1994-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Survival time | 22 years

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Sirikit Centre for Breast Cancer, Bangkok, Bangkok, Thailand